CLINICAL TRIAL: NCT01033877
Title: Immunogenicity and Safety of a Tetanus, Diphtheria and Mono Component Acellular Pertussis (TdaP) Vaccine in Comparison to a Tetanus and Diphtheria (Td) Vaccine When Given as a Booster Vaccination to Adults
Brief Title: Immunogenicity and Safety of Tetanus, Diphtheria and Mono Component Acellular Pertussis (TdaP) Vaccine in Comparison to Tetanus and Diphtheria (Td) Vaccine When Given as Booster Vaccinations to Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VTdaP-01
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: Immunisation, active
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TdaP vaccine (Experimental)
  Interventions: Biological: TdaP vaccine SSI
- Td vaccine (Active Comparator)
  Interventions: Biological: Td vaccine SSI

INTERVENTIONS:
Biological: TdaP vaccine SSI — 1 vaccine dose of 0.5 mL suspension for injection in a pre-filled syringe: >= 20 I.U. tetanus toxoid (T), >=2 I.U. diphtheria toxoid (d), 20 microgram pertussis toxoid (aP)
  Arms: TdaP vaccine
Biological: Td vaccine SSI — 1 vaccine dose of 0.5 mL suspension for injection in a pre-filled syringe: >= 20 I.U. tetanus toxoid (T), >=2 I.U. diphtheria toxoid (d)
  Arms: Td vaccine

SUMMARY:
The clinical trial is a phase III, double-blind, randomised, controlled, multi-centre, clinical trial, on the immunogenicity and safety of TdaP vaccine in comparison to Td vaccine when given as a booster vaccination to adults who were vaccinated with D, T and wP vaccine according to the Danish vaccination programme in their childhood.

Healthy, adult, female or male volunteers, who completed primary vaccination with diphtheria (D), tetanus (T) and whole cell pertussis vaccine (wP), typically during their childhood, is the target population.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female or male adult of ≥ 18 years of age
2. Completed primary vaccination with diphtheria (D), Tetanus (T) and whole cell pertussis (wP) vaccines in Denmark
3. Signed informed consent
4. Prepared to grant authorised persons access to medical records
5. Likely to comply with instructions

Exclusion Criteria:

1. Congenital or acquired immunodeficiency or progressive neurologic disease
2. Uncontrolled epilepsy or progressive encephalopathy
3. Previous experience of serious adverse reaction(s) after vaccinations with diphtheria-, tetanus- acellular or whole cell pertussis- vaccines
4. Vaccinated with any diphtheria, tetanus or pertussis toxoid containing vaccine within 5 years before inclusion
5. Vaccinated with any tetanus toxoid, diphtheria toxoid or diphtheria CRM197 protein conjugated vaccine within 5 years before inclusion
6. Known tetanus-, diphtheria- or pertussis disease/infection within 5 years before inclusion
7. Known hypersensitivity or history of allergic reactions to any of the active or inactive constituents of the TdaP or Td vaccines
8. Vaccinated with a live or inactivated vaccine within 1 month before inclusion
9. Administration of immune modulating drugs (such as immunoglobulin, systemic corticosteroids, blood products, azathioprine, cyclosporine, infliximab) within 3 months before inclusion
10. Administration of any investigational drug product or vaccine within 1 month before inclusion
11. Females if pregnant or breastfeeding or not willing to use contraception during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 802 (Actual)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Three co-primary outcome measures: Serum anti-PTx antibody conc. in pre- and post-vac. serum samples | one month post-vaccination
Serum anti-diphtheria antibody conc. in post-vac. serum samples | one month post -vaccination
Serum anti-tetanus antibody conc. in post-vac. serum samples | one month post-vaccination

SECONDARY OUTCOMES:
Three secondary outcome measures: Local and systemic adverse events reported during one month following the vaccination | one month post-vaccination
Serum anti-diphtheria antibody conc. in pre-vac. serum samples | one month post-vaccination
Serum anti-tetanus antibody conc. in pre-vac. serum samples | one month post- vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Thierry-Carstensen, M.Sc. Pharm, Study Director — Statens Serum Institut; Carsten Heilmann, Professor MD, Principal Investigator — H:S Rigshospitalet
Locations (2):
- Denmark (2):
  - H:S Rigshospitalet, Copenhagen
  - aCROnordic, Hoersholm

REFERENCES:
- [Derived] Thierry-Carstensen B, Jordan K, Uhlving HH, Dalby T, Sorensen C, Jensen AM, Heilmann C. A randomised, double-blind, non-inferiority clinical trial on the safety and immunogenicity of a tetanus, diphtheria and monocomponent acellular pertussis (TdaP) vaccine in comparison to a tetanus and diphtheria (Td) vaccine when given as booster vaccinations to healthy adults. Vaccine. 2012 Aug 10;30(37):5464-71. doi: 10.1016/j.vaccine.2012.06.073. Epub 2012 Jul 6. PMID 22776216